CLINICAL TRIAL: NCT03102879
Title: Encapsulated Mesenchymal Stem Cells for Endodontic Treatment of Permanent Teeth With Apical Lesion: a Controlled Clinical Trial.
Brief Title: Encapsulated Mesenchymal Stem Cells for Dental Pulp Regeneration.
Acronym: RanoKure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Cells for Cells (Industry)
Responsible Party: Principal Investigator, Dra. Claudia Brizuel, Doctor of Dental Surgery, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RPD-8-16
Record Dates: First submitted 2017-03-21; First posted 2017-04-06 (Actual); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Periapical Periodontitis
Keywords: mesenchymal stem cells; regenerative procedures; tissue engineering; regenerative endodontic; scaffold; cell encapsulation; dental pulp; pulp regeneration; plasma-derived biomaterial; allogenic stem cells; mesenchymal stromal cells; adult stem cells; umbilical cord stem cells
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: 2 interventions:
  1. Endodontic regenerative treatment with Biological product of umbilical cord-derived mesenchymal stem cells encapsulated in a plasma-derived biomaterial.
  2. Endodontic treatment with inert product gutapercha.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regenerative Endodontic Procedure (REP) (Experimental): umbilical cord-derived mesenchymal stem cells encapsulated in a plasma-derived biomaterial.
  Interventions: Procedure: Regenerative Endodontic Procedure
- Conventional Root Canal Treatment (Active Comparator): Conventional endodontic procedure
  Interventions: Procedure: Conventional Root Canal Treatment

INTERVENTIONS:
Procedure: Regenerative Endodontic Procedure — Coronary access, conductometry, mechanized instrumentation, irrigation with sodium hypochlorite, intracanal calcium hydroxide medication and obturation with stem cells.
  Other Names: REP; Tissue engineering procedure
  Arms: Regenerative Endodontic Procedure (REP)
Procedure: Conventional Root Canal Treatment — Coronary access, conductometry, mechanized instrumentation, irrigation with sodium hypochlorite, intracanal calcium hydroxide medication and obturation with gutta-percha.
  Other Names: Gold standard treatment
  Arms: Conventional Root Canal Treatment

SUMMARY:
To compare the dental survival in a period of one year of mature permanent teeth with apical lesion following the administration of encapsulated Mesenchymal Stem Cells under a regenerative endodontic procedure and a conventional root canal treatment.

DETAILED DESCRIPTION:
This is a controlled clinical trial designed to evaluate the survival of mature permanent teeth with apical lesion treated with regenerative endodontic procedure (REP) based on encapsulated Mesenchymal Stem Cells in a biological scaffold. The REP will be compared to the conventional endodontic therapy. The REP is based on the use of umbilical cord-derived mesenchymal stem cells encapsulated in a plasma-derived biomaterial . The study group will use the disinfection protocol, indicated in the clinical considerations for regenerative procedures as recommended by the American Association of Endodontics, using a paste of calcium hydroxide prepared with double-distilled water as intracanal medication, and will be operated with REP using allogeneic stem cells in a scaffold, while the control group will be operated with conventional endodontic therapy alone. This clinical trial pretends to determine the dental survival of the tooth with mature apex and apical lesion, over a period of one year.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria:

* Age: 16 - 58 years old.
* Signed the informed consent.
* Non-smoking.
* Systemically healthy patients

Tooth inclusion criteria:

* Upper and lower incisors, upper and lower canines and lower premolars teeth with mature apex and apical lesion (greater than 2 PAI and 1 CBCTPAI).
* Teeth that do not response to both electrical and thermal pulp test
* Teeth that can be restored (as defined by Class A or Class B using Samet and Jotkowitz classification) without the need of a stainless steel crown.

Exclusion Criteria:

Patient exclusion criteria:

* Patients without a phone number for contact during the study.
* Subjects not available for follow up period (12 months).
* Patients who are or will undergo orthodontic treatment over the next 12 months.
* Patients with an allergy to any material or drug used in the study.
* Patients who are pregnant or lactating.
* Patients with a history of systemic diseases that alter immune function, such as diabetes mellitus, immunodeficiency, leukemia, Addison's disease and Cushing.
* Patients who have used immunosuppressive drugs or chemotherapy, 3 months before the study.

Tooth exclusion criteria:

* Endodontically treated teeth
* Teeth with signs of severe root resorption.
* Teeth with mobility class III or Dens invaginatus.
* Teeth with avulsion history and conservation in a dry extraoral medium for more than 1 hour.
* Teeth with clinical and / or radiographic evidence of root fracture.
* Teeth that can not be absolutely isolated with rubber dam. . Teeth with more than one root or root canal.

Ages: 16 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brizuela C, Meza G, Urrejola D, Quezada MA, Concha G, Ramirez V, Angelopoulos I, Cadiz MI, Tapia-Limonchi R, Khoury M. Cell-Based Regenerative Endodontics for Treatment of Periapical Lesions: A Randomized, Controlled Phase I/II Clinical Trial. J Dent Res. 2020 May;99(5):523-529. doi: 10.1177/0022034520913242. Epub 2020 Mar 23. PMID 32202965

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between September 2016 and September 2017, from patients referred for endodontic treatment to the Universidad de los Andes Health Center, located in San Bernardo city, Santiago, Chile.
Groups:
- Regenerative Procedure: Endodontic regenerative treatment with Biological product of umbilical cord-derived mesenchymal stem cells encapsulated in a plasma-derived biomaterial.
- Endodontic Treatment: Conventional root canal treatment treatment with inert product gutapercha.
Period: Overall Study
Arm/Group | Regenerative Procedure | Endodontic Treatment
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regenerative Procedure | Endodontic Treatment | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 27 [22 to 39] | 28 [24 to 43] | 27 [23 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participats Showing Efficacy (Functionality)
Description: Efficacy (functionality) was defined when one year after the intervention, the treated tooth remains in the mouth, without pain to percussion test and with apical bone lesion of equal size in the three senses of space or a decrease in some of them or no more than 0.1 mm increase of one of them.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Regenerative Procedure | Endodontic Treatment
Number analyzed (Participants) | 18 | 18
Participants | 18 | 18

2. Secondary Outcome: Change in Pulpal Response
Description: Change in pulpal response (period 1 year) will be assessed through response to sensitivity tests (cold, hot and electrical test) in teeth treated with regenerative procedure and conventional endodontic treatment during time.
Time Frame: baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Conventional Treatment: Conventional Endodontic treatment
Arm/Group | Regenerative Procedure | Conventional Treatment
Number analyzed (Participants) | 18 | 18
Participants
  Basal Cold Test: Response | 1 | 1
  Basal Cold Test: No Response | 17 | 17
  Basal Hot Test: Response | 0 | 1
  Basal Hot Test: No Response | 18 | 17
  Basal Electrical Test: Response | 3 | 1
  Basal Electrical Test: No Response | 15 | 17
  6 months Cold Test: Response | 14 | 2
  6 months Cold Test: No Response | 4 | 16
  6 months Hot Test: Response | 2 | 0
  6 months Hot Test: No Response | 16 | 18
  6 months Electrical Test: Response | 4 | 4
  6 months Electrical Test: No Response | 14 | 14
  12 months Cold Test: Response | 10 | 1
  12 months Cold Test: No Response | 8 | 17
  12 months Hot Test: Response | 5 | 0
  12 months Hot Test: No Response | 13 | 18
  12 months Electrical Test: Response | 9 | 3
  12 months Electrical Test: No Response | 9 | 15

3. Secondary Outcome: Change in Apical Lesion Size
Description: Change in apical lesion size will be evaluated by cone beam tomography 6 and 12 months after intervention is completed.
Time Frame: baseline, 6 months, 12 months
Measure: Median (Inter-Quartile Range); unit: milimeters
Arm/Group | Regenerative Endodontic Procedure (REP) | Conventional Root Canal Treatment
Number analyzed (Participants) | 18 | 18
milimeters
  Basal Mesio-Distal | 5 [4.2 to 7.7] | 5.5 [3.3 to 6.7]
  Basal Height | 5.5 [4.7 to 8.9] | 7.1 [2.9 to 10.1]
  Basal Antero-Posterior | 5 [4.6 to 6] | 5.1 [3.3 to 6.2]
  6 months Mesio-Distal | 2.7 [2 to 5.1] | 2.4 [0.9 to 5.9]
  6 months Height | 2.6 [2.4 to 4.6] | 2.5 [1.4 to 4.3]
  6 months Antero-Posterior | 2.4 [2.2 to 4.4] | 3 [1.7 to 4]
  12 months Mesio-Distal | 2 [1.4 to 3.4] | 1.7 [0.9 to 3.4]
  12 months Height | 1.8 [0.8 to 4.1] | 1.5 [0.4 to 4.4]
  12 months Anterio-Posterior | 2.1 [1.1 to 4.1] | 1.7 [0.6 to 3.3]

4. Secondary Outcome: Pain to Percussion
Description: To compare pain to percussion in a period of 1 year in permanent teeth with mature apex and apical lesion, treated with a regenerative endodontic procedure and conventional endodontic therapy.
  This will be monitored 6 and 12 months after the procedure is completed.
  Pain to percussion positive: The tooth is tenderness when is softly tapped with handle end of a dental mirror at examination time.
  Pain to percussion negative: The tooth is not tenderness when is softly tapped with handle end of a dental mirror at examination time.
Time Frame: baseline, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Regenerative Procedure | Conventional Treatment
Number analyzed (Participants) | 18 | 18
Participants
  Baseline Pain to Percussion: Positive | 11 | 5
  Baseline Pain to Percussion: Negative | 7 | 13
  6 months Pain to Percussion: Positive | 1 | 0
  6 months Pain to Percussion: Negative | 17 | 18
  12 months Pain to Percussion: Positive | 0 | 0
  12 months Pain to Percussion: Negative | 18 | 18

5. Secondary Outcome: Numbers of Participants With Adverse Event
Description: To describe adverse events in a period of 1 year in permanent teeth with mature apex and apical lesion, operated with a regenerative endodontic procedure and conventional endodontic therapy.
Time Frame: 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Regenerative Procedure | Conventional Treatment
Number analyzed (Participants) | 18 | 18
Participants
  6 months | 0 | 0
  12 months | 0 | 0

6. Secondary Outcome: Pulp Regeneration
Description: To describe the pulp regeneration by means of vitality test using Doppler laser flowmetry (LDF) in a period of 1 year in permanent teeth with mature apex and apical lesion treated with a regenerative endodontic procedure.
  The vitality of the teeth was measured by LDF and the perfusion units (PU) percentage of the tooth under study was determined with respect to a healthy control tooth with similar anatomical characteristics from the same patient.
Time Frame: baseline, 6 months, 12 months
Population: This outcome was not measured in conventional treatment group due to the nature of the filling material, which does not promote revitalization of the pulp.
Measure: Median (Inter-Quartile Range); unit: % PU in time in relation to controltooth
Arm/Group | Regenerative Procedure
Number analyzed (Participants) | 18
% PU in time in relation to controltooth
  Basal | 60.6 [53.5 to 75]
  6 months | 74.4 [49.2 to 102.2]
  12 months | 78.1 [54.7 to 99.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a period of 1 year in permanent teeth with mature apex and apical lesion, operated with a regenerative endodontic procedure and conventional endodontic therapy.
Description: Safety encompassed immediate adverse events after implantation of UC-MSCs in the REP group or gutta-percha in the ENDO group, as defined by root fracture, severe or moderate pain and extra-intraoral inflammation.
Arm/Group | Regenerative Procedure | Conventional Treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03102879/Prot_SAP_000.pdf